CLINICAL TRIAL: NCT00438022
Title: Risk Factors in Atopic Dermatitis for the Development of Eczema Herpeticum
Brief Title: Identifying Risk Factors for Eczema Herpeticum in Individuals With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis and Vaccinia Network (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ADVN ADEH 06; HHSN266200400029C (Other: NIH Contract)
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Atopic Dermatitis; Eczema Herpeticum
Keywords: Atopic Dermatitis; Eczema Herpeticum
MeSH Terms: conditions — Dermatitis, Atopic; Kaposi Varicelliform Eruption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and skin samples will be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Group 1 will include participants with AD, EH, and recurrent herpes simplex virus (HSV)
- 2: Group 2 will include participants with AD and recurring HSV infections but without EH
- 3: Group 3 will include participants with AD but without EH or HSV infection
- 4: Group 4 will include participants in good general health without AD, EH, or HSV infection

SUMMARY:
Atopic Dermatitis (AD), also known as eczema, is a skin disease that causes the skin to be hot, dry and scaly, and have severe itching. There are different kinds of eczema. Eczema herpeticum (EH) is a type of eczema that spreads due to an underlying herpes virus infection. The purpose of this research study is to identify the risk factors that may cause EH.

DETAILED DESCRIPTION:
AD is characterized by chronic skin inflammation and infections. It is hypothesized that AD is caused by irritants in the environment and that symptoms of EH become worse with stress and changes in hormone levels. This study will examine skin cells collected from study participants to determine the risk factors for EH that are present in people with AD who develop EH.

This study will examine dendritic cells (DC) from the skin and blood of study participants to determine the differences between DCs of study participants. This study will recruit four types of participants:

* Group 1 will include participants with AD, EH, and recurrent herpes simplex virus (HSV)
* Group 2 will include participants with AD and recurring HSV infections but without EH
* Group 3 will include participants with AD but without EH or HSV infection
* Group 4 will include participants in good general health without AD, EH, or HSV infection

At the single study visit, skin and blood collection will occur.

ELIGIBILITY:
Inclusion Criteria for Participants with AD:

* Diagnosis of AD as defined by ADVN standardized diagnostic criteria who fall into one of the following categories:

  1. Recurrent, clinically manifested HSV infection with EH
  2. Recurrent, clinically manifested HSV infection without EH
  3. No recurrent, clinically manifested HSV infection or EH infection

Inclusion Criteria for All Participants

* Residing in Germany
* Good general health other than having an atopic disease
* Caucasian
* Individuals between 18-60 years of age

Exclusion Criteria for All Participants:

* Subjects with atopy but lacking stringent AD features, allowing only a presumptive diagnosis of AD
* Individuals under 18 or over 60 years of age
* Systemic immunosuppressive drugs or chemotherapy 30 days prior to study entry
* Oral and topical corticosteroids (including inhaled agents), antibiotics, antivirals, anti-inflammatory biologics (e.g., alefacept, etanercept), topical doxepin, topical coal tar preparations, or topical phosphodiesterase inhibitors 14 days prior to study entry
* Immunotherapy
* Antibiotics, antivirals, immune enhancers (e.g., imiquimod), or calcineurin inhibitors within 7 days prior to study entry
* Phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA]) 30 days prior to study entry
* Cancer, autoimmune diseases, or immunodeficiency
* Active fungal, bacterial, or viral infections at screening
* Any skin diseases other than AD that might compromise the stratum corneum barrier (e.g., ichthyosis, bullous disease, psoriasis, skin cancer)
* Mental illness or a history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
* Inability or unwillingness of a subject to give written informed consent
* Weigh less than 40 kg (88.2 lb)
* Anxiolytic agents
* Antidepressants
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People of good general health, living in Germany
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Immunohistochemistry will be used to confirm the expression of IgE receptors and IgE binding of myeloid and plasmacytoid Dendritic Cells. | 3 years

SECONDARY OUTCOMES:
The capacity of myeloid and plasmacytoid DCs to produce IFN-α/IFN-β and of myeloid DCs to produce IL-10, IL-12, and IL-18 will be evaluated. | 3 years
Expression of HSV-receptors cluster of differentiation, costimulatory molecules, major histocompatibility complex, Toll-like receptor (TLR), and structures involved in antigen presentation of myeloid and plasmacytoid DCs. | 3 years
Evaluate the capacity of T-cells, stimulated and unstimulated myeloid DCs or plasmacytoid DCs to produce the T-helper cell 2 (Th2) cytokines IL-4, IL-5 and IL-13 and the T-helper cell 1 (Th1) cytokines IL-2 and IFN-γ and IL-10/TGF-β. | 3 years
The phenotype of T-cells cocultured with HSV/CpG stimulated and unstimulated myeloid DCs or plasmacytoid DCs will be evaluated by flow cytometry. | 3 years
The proliferation of T-cells cocultured with HSV/CpG stimulated and unstimulated myeloid DCs or plasmacytoid DCs will be measured with the help of flow cytometry by proliferating cell nuclear antigen. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bieber, MD, PhD, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Germany, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access is available to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Peng WM, Yu CF, Allam JP, Oldenburg J, Bieber T, Hoch J, Eis-Hubinger AM, Novak N. Inhibitory oligodeoxynucleotides downregulate herpes simplex virus-induced plasmacytoid dendritic cell type I interferon production and modulate cell function. Hum Immunol. 2007 Nov;68(11):879-87. doi: 10.1016/j.humimm.2007.10.008. Epub 2007 Nov 5. PMID 18082566
- [Result] Hinz T, Zaccaro D, Byron M, Brendes K, Krieg T, Novak N, Bieber T. Atopic dermo-respiratory syndrome is a correlate of eczema herpeticum. Allergy. 2011 Jul;66(7):925-33. doi: 10.1111/j.1398-9995.2010.02538.x. Epub 2011 Jan 24. PMID 21255038
- See also: National Institute of Allergy and Infectious Diseases (NIAID) Website — https://www.niaid.nih.gov/research/role
- Available data/document: Individual Participant Data Set: Study ID is SDY4 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY4
- Available data/document: Study Protocol: Study ID is SDY4 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY4
- Available data/document: Study details, -download packages, et al.: Study ID is SDY4 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY4